CLINICAL TRIAL: NCT03660462
Title: Iron Bioavailability of High Surface Area Ferric Phosphate in Thai Women
Brief Title: Iron Bioavailability of High Surface Area Ferric Phosphate
Acronym: HiFe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr. med., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HiFe
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FeSO4 fortified rice test meal (Active Comparator)
  Interventions: Dietary Supplement: FeSO4 fortified rice test meal
- FePO4 fortified rice test meal (Experimental)
  Interventions: Dietary Supplement: FePO4 fortified rice test meal
- HiFePO4 1 fortified rice test meal (Experimental)
  Interventions: Dietary Supplement: HiFePO4 1 fortified rice test meal
- HiFePO4 2 fortified rice test meal (Experimental)
  Interventions: Dietary Supplement: HiFePO4 2 fortified rice test meal

INTERVENTIONS:
Dietary Supplement: FeSO4 fortified rice test meal — Rice test meal extrinsically labeled with 2 mg ferrous sulfate (58FeSO4)
  Arms: FeSO4 fortified rice test meal
Dietary Supplement: FePO4 fortified rice test meal — Rice test meal extrinsically labeled with 2 mg ferric phosphate (58FePO4)
  Arms: FePO4 fortified rice test meal
Dietary Supplement: HiFePO4 1 fortified rice test meal — Rice test meal extrinsically labeled with 2 mg high surface ferric phosphate 1 (57FePO4)
  Arms: HiFePO4 1 fortified rice test meal
Dietary Supplement: HiFePO4 2 fortified rice test meal — Rice test meal extrinsically labeled with 2 mg high surface ferric phosphate 2 (57FePO4)
  Arms: HiFePO4 2 fortified rice test meal

SUMMARY:
The primary objective of this study is to compare iron absorption of high surface area ferric phosphate with that of ferrous sulfate and bulk ferric phosphate in a rice-based meal in non-pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (18 to 49 years) in Thailand
* BMI < 23 kg/m2
* Body weight < 65 kg
* Mildly anaemic to normocythemic (Hb 80-110 g/L)
* Ferritin < 25 µg/L
* Not pregnant (confirmed by pregnancy test stripe) or lactating
* No inflammation (CRP < 5 mg/L)
* Having provided written informed consent

Exclusion Criteria:

* Haemoglobinopathies (except heterozygosity for haemoglobin E and alpha-thalassemia 1)
* Coeliac disease or other chronic diseases of malabsorption that could influence iron absorption or metabolism
* Blood donation or significant blood loss due to surgery or accident < 4 months before start of the study
* Consumption of vitamin or mineral supplements 2 weeks before start of the study
* Regular use of medication (except oral contraceptives), that influences iron absorption
* Chronic inflammatory disease
* Smoking

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption | Measured 14 days after consumption of the 4 different types of iron vehicles (Days 16 and 31)
  Iron absorption will be determined by measurement of the isotopic ratio change from the 4 different types of iron vehicles (FeSO4 fortified rice test meal, FePO4 fortified rice test meal, HiFePO4 1 fortified rice test meal, HiFePO4 2 fortified rice test meal).

CONTACTS AND LOCATIONS:
Locations (1):
- Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No